CLINICAL TRIAL: NCT04859634
Title: Real-time Artificial Intelligence System for Detecting Multiple Ocular Fundus Lesions by Ultra-widefield Fundus Imaging: A Prospective Multicenter Study
Brief Title: Real-time Artificial Intelligence System for Detecting Multiple Ocular Fundus Lesions by Ultra-widefield Fundus Imaging
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Shenzhen Eye Hospital (Other); Xudong Ophthalmic Hospital (Unknown); IKang Physical Examination Center (Unknown); Beijing Tongren Hospital (Other); Guangdong Provincial People's Hospital (Other); Yangxi General Hospital People's Hospital (Unknown)
Responsible Party: Principal Investigator, Haotian Lin, Professor, Sun Yat-sen University
Other Study IDs: UWFAIDS2019-China-06
Record Dates: First submitted 2021-04-15; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Artificial Intelligence; Diagnostic Imaging; Abnormality of the Fundus; Diagnostic Screening Programs
Keywords: Artificial Intelligence; Deep learning; Ultra-widefield Fundus Imaging; Ocular Fundus Lesions; Diagnostic Screening Programs

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (7):
- Zhongshan Ophthalmic Center: The participant only needs to take an ultra-widefield fundus image as usual.
  Interventions: Device: Taking an ultra-widefield fundus image
- Shenzhen Ophthalmic Center: The participant only needs to take an ultra-widefield fundus image as usual.
  Interventions: Device: Taking an ultra-widefield fundus image
- Beijin Tongren Hospital: The participant only needs to take an ultra-widefield fundus image as usual.
  Interventions: Device: Taking an ultra-widefield fundus image
- Xudong Ophthalmic Center: The participant only needs to take an ultra-widefield fundus image as usual.
  Interventions: Device: Taking an ultra-widefield fundus image
- IKang Physical Examination Center: The participant only needs to take an ultra-widefield fundus image as usual.
  Interventions: Device: Taking an ultra-widefield fundus image
- Yangxi General Hospital People's Hospital: The participant only needs to take an ultra-widefield fundus image as usual.
  Interventions: Device: Taking an ultra-widefield fundus image
- Guangdong Provincial People's Hospital: The participant only needs to take an ultra-widefield fundus image as usual.
  Interventions: Device: Taking an ultra-widefield fundus image

INTERVENTIONS:
Device: Taking an ultra-widefield fundus image — The participant only needs to take an ultra-widefield fundus image as usual.

SUMMARY:
This prospective multicenter study will evaluate the efficacy of a real-time artificial intelligence system for detecting multiple ocular fundus lesions by ultra-widefield fundus imaging in real-world settings.

DETAILED DESCRIPTION:
The ocular fundus can show signs of both ocular diseases (e.g., lattice degeneration, retinal detachment and glaucoma) and systemic diseases (e.g., hypertension, diabetes and leukemia). The routine fundus examination is conducive for early detection of these diseases. However, manual conducting fundus examination needs an experienced retina ophthalmologist, and is time-consuming and labor-intensive, which is difficult for its routine implementation on large scale.

This study will develop an artificial intelligence system integrating with ultra-widefield fundus imaging to automatically screen for multiple ocular fundus lesions in real time and evaluate its performance in different real-world settings. The efficacy of the system will compare to the final diagnoses of each participant made by experienced ophthalmologists.

ELIGIBILITY:
Inclusion Criteria:

All the participants who agree to take ultra-widefield fundus images.

Exclusion Criteria:

1. Patients who cannot cooperate with a photographer such as some paralytics, the patients with dementia and severe psychopaths.
2. Patients who do not agree to sign informed consent.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All the participants who agree to take ultra-widefield fundus images.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-12-25 (Estimated)

PRIMARY OUTCOMES:
Accuracy | 8 months
  Performance of artificial intelligence system for detecting multiple ocular fundus lesions based on ultra-widefield fundus imaging.

SECONDARY OUTCOMES:
Sensitivity | 8 months
  Performance of artificial intelligence system for detecting multiple ocular fundus lesions based on ultra-widefield fundus imaging.
Specificity | 8 months
  Performance of artificial intelligence system for detecting multiple ocular fundus lesions based on ultra-widefield fundus imaging.
Cohen's kappa coefficient | 8 months
  The comparison between the performacne of AI system and ophthalmologists of three degrees of expertise.
False-positive rate | 8 months
  Features of Misclassification
False-negative rate | 8 months
  Features of Misclassification
Data processing time of AI system | 8 months
  Data processing time of AI system.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China